CLINICAL TRIAL: NCT00507273
Title: Gastrointestinal Stromal Tumors (GIST) Registry Protocol: reGISTry
Brief Title: Gastrointestinal Stromal Tumors (GIST) Registry
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 2005-0294
Record Dates: First submitted 2007-07-25; First posted 2007-07-26 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; Gastrointestinal Cancer; GISTs; GIST Registry; Registry
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- GIST: Patients diagnosed with a gastrointestinal stromal tumor (GIST)
  Interventions: Other: GIST Registry

INTERVENTIONS:
Other: GIST Registry — Internet based data registry about how different physicians treat and manage patients with gastrointestinal stromal tumors.

SUMMARY:
The goal of this observational research study is to establish a registry of information regarding how different physicians treat and manage patients with gastrointestinal stromal tumors (GISTs).

Objectives:

1. To describe variation in management of patients with GIST, overall and by patient and provider characteristics.
2. To provide participating physicians with information regarding management of their patients with GIST compared to the aggregate experience of all physicians participating in the Registry.

DETAILED DESCRIPTION:
The Registry, which is Internet based, is intended to collect information about current practices in the management of GIST without making any specific change to the standard of care as decided by each patient's treating physician.

If you agree to participate in this study, your doctor will provide information to a data registry about your physical and clinical traits, the past and current medical care you have received to treat your GIST, and clinically-related, economically-related, and health-related quality of life information. About 200 doctors will provide information on their patients for the Registry. Your doctor will collect this information when you first join the Registry and at each regularly scheduled visit you make to your doctor's office. The information collection will continue for as long as you and your doctor feel it is appropriate. The information that is entered into the Registry will remain there indefinitely. It is hoped that this sharing of information will lead to a better understanding of how to best treat patients with GIST.

You and your doctor will decide what treatment you will receive. Because this Registry is only to observe actual medical practice, it does not require you to receive any particular treatment.

Only your doctor and people who will help your doctor collect the information for this Registry will know which information submitted to the Registry belongs to you. Data will be tracked in the Registry using only ID numbers and patient initials. The information submitted on the Registry data collection forms will not be associated with a specific patient's identity. Separately, you will be asked to provide your name, place of birth, and Social Security number. This information will not be entered into the Registry databases and will only be used if it is necessary to perform a search should you become lost to follow up. If you do not want to provide your Social Security number you may still be enrolled in the Registry.

This is an investigational study. About 100 patients from M. D. Anderson will be entered into the Registry. In all, about 1800 patients will be registered. The Registry will be active for at least 7 years.

ELIGIBILITY:
Inclusion Criteria:

1. All patients who have been diagnosed with GIST are eligible for enrollment.

Exclusion Criteria:

1. Patients with a histologic diagnosis other than gastrointestinal stromal tumor (GIST).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with a gastrointestinal stromal tumor (GIST).
Sampling Method: Non-Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2005-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Current patterns of medical practice in management of patients with GIS | 5 Years
  Data from observational GIST Registry analyzed to describe current patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Trent, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pisters PWT, Blanke CD, von Mehren M, Picus J, Sirulnik A, Stealey E, Trent JC; reGISTry Steering Committee. A USA registry of gastrointestinal stromal tumor patients: changes in practice over time and differences between community and academic practices. Ann Oncol. 2011 Nov;22(11):2523-2529. doi: 10.1093/annonc/mdq773. Epub 2011 Apr 4. PMID 21464155
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org